CLINICAL TRIAL: NCT00708162
Title: A Multicenter, Randomized, Double-Blind, Double-Dummy, Phase 3 Study of the Safety and Efficacy of Ritonavir-Boosted Elvitegravir (EVG/r) Versus Raltegravir (RAL) Each Administered With a Background Regimen in HIV-1 Infected, Antiretroviral Treatment-Experienced Adults
Brief Title: Multicenter, Randomized, Double-Blind, Double-Dummy, Phase 3 Study of the Safety and Efficacy of Elvitegravir Versus Raltegravir
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GS-US-183-0145; 2007-004225-26 (EudraCT Number); NCT00707733 (obsolete NCT alias)
Record Dates: First submitted 2008-06-30; First posted 2008-07-02 (Estimated); Results first posted 2014-11-06 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-04

CONDITIONS: HIV Infection
Keywords: HIV; HIV I; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — elvitegravir; Raltegravir Potassium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Elvitegravir (Experimental): EVG 85 mg or 150 mg + RAL placebo + background regimen in the Randomized Phase, followed by EVG 85 mg or 150 mg + background regimen in the Open-Label Phase.
  Participants receiving lopinavir/ritonavir (LPV/r) or atazanavir/ritonavir (ATV/r) as part of their background regimen will receive EVG 85 mg; all other participants will receive EVG 150 mg.
  Interventions: Drug: Elvitegravir; Drug: RAL placebo; Drug: Background regimen
- Raltegravir (Active Comparator): RAL 800 mg (400 mg twice daily) + EVG placebo + background regimen in the Randomized Phase, followed by EVG 85 mg or 150 mg + background regimen in the Open-Label Phase.
  Participants receiving LPV/r or ATV/r as part of their background regimen in the Open-Label Phase will receive EVG 85 mg; all other participants will receive EVG 150 mg.
  Interventions: Drug: Raltegravir; Drug: EVG placebo; Drug: Background regimen

INTERVENTIONS:
Drug: Elvitegravir — Elvitegravir (EVG) tablet administered orally once daily with food
  Other Names: Vitekta®; GS-9137
  Arms: Elvitegravir
Drug: Raltegravir — Raltegravir tablet administered orally twice daily according to prescribing information
  Other Names: Isentress®
  Arms: Raltegravir
Drug: EVG placebo — Placebo to match elvitegravir administered orally once daily
  Arms: Raltegravir
Drug: RAL placebo — RAL placebo administered orally twice daily.
  Arms: Elvitegravir
Drug: Background regimen — Background Regimen (administered according to prescribing information) contains 1 fully-active ritonavir-boosted protease inhibitor (PI/r) plus 1 or 2 additional agents. The ritonavir-boosted PIs include either ATV, darunavir, fosamprenavir, LPV (Kaletra®), or tipranavir; the additional agents include abacavir (ABC), Combivir® (lamivudine (LAM)/zidovudine (ZDV) coformulated), didanosine, emtricitabine (FTC), enfuvirtide, Epzicom® (ABC/LAM coformulated), etravirine, LAM, maraviroc, tenofovir disoproxil fumarate (TDF), Truvada®, (FTC/TDF coformulated), and/or ZDV.

SUMMARY:
The purpose of this study is to compare the safety, tolerability and efficacy of a regimen containing once-daily elvitegravir (EVG) versus twice-daily raltegravir (RAL) added to a background regimen (1 fully-active ritonavir (RTV)-boosted protease inhibitor (PI) plus 1 or 2 additional antiretroviral (ARV) agents) in HIV-1 infected, ARV treatment-experienced adults who have documented resistance, or at least six months experience prior to screening with two or more different classes of ARV agents.

Participants will be randomized in a 1:1 ratio to receive EVG plus background regimen (Elvitegravir group), or raltegravir plus background regimen (Raltegravir group). Due to known drug interactions, participants in the Elvitegravir group receiving RTV-boosted atazanavir (ATV) or RTV-boosted lopinavir (LPV) as part of their background regimen will receive elvitegravir at a lower dose (85 mg).

DETAILED DESCRIPTION:
The background regimen will be constructed by the investigator based on viral resistance testing. The fully active PI will be defined by phenotypic resistance analysis. For phenotypic susceptibility, fully active is defined as being below the lower clinical or biological cutoff. Participants are required to take their ritonavir dose based on the dosing schedule indicated in the prescribing information for the PI; no additional ritonavir is required to be taken with EVG. No other marketed PIs are allowed as part of the background regimen due to unknown drug interactions.

The second agent can be one nucleoside or nucleotide reverse transcriptase inhibitor (NRTI), etravirine, maraviroc, or T-20. However, the second agent must not include an integrase inhibitor; the nonnucleoside reverse transcriptase inhibitors efavirenz, nevirapine, or delavirdine (due to unknown drug interactions); or the fixed-dose combination therapies Atripla® or Trizivir® (abacavir sulfate/lamivudine/zidovudine). The second agent may or may not be fully active (except in Spain, where participants have to receive a fully active second agent, as requested by the Spanish regulatory agency).

If the M184V/I reverse transcriptase (RT) mutation is present on the screening genotype report and an NRTI is used as the second agent, then either FTC or LAM may be added as a third agent in the background regimen to maintain the M184V/I mutation. In this situation only, the fixed-dose combination therapies Combivir®, Truvada®, or Epzicom/Kivexa® may be prescribed as the combined second and third agents of the background regimen.

After Week 96, participants will continue to take their blinded study drug and attend visits until treatment assignments are unblinded, at which point they will be given the option to participate in an open-label EVG extension phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* Plasma HIV-1 RNA levels ≥ 1,000 copies/mL at screening
* Documented resistance or at least six months experience prior to screening with two or more different classes of antiretroviral agents
* Stable antiretroviral regimen for at least 30 days prior to screening: however, participants may discontinue the antiretroviral regimen after screening and remain off therapy until baseline at the discretion of the investigator
* Eligible to receive one of the fully-active ritonavir-boosted-PIs, and an allowed second agent
* Normal ECG
* Adequate renal function (estimated glomerular filtration rate according to the Cockcroft-Gault formula ≥ 60 mL/min)
* Hepatic transaminases ≤ 5 × upper limit of normal
* Total bilirubin ≤ 1.5 mg/dL, or normal direct bilirubin
* Adequate hematologic function (absolute neutrophil count ≥ 1,000/mm^3; platelets ≥ 50,000/mm^3; hemoglobin ≥ 8.5 g/dL)
* Serum amylase < 1.5 × the upper limit of the normal range
* Negative serum pregnancy test (females of childbearing potential only)
* Males and females of childbearing potential must agree to use highly effective contraception methods
* Age ≥ 18 years
* Life expectancy ≥ 1 year
* Ability to understand and sign a written informed consent form

Exclusion Criteria:

* New AIDS-defining condition diagnosed within the 30 days prior to screening
* Prior treatment with any HIV-1 integrase inhibitor
* Participants experiencing ascites
* Participants experiencing encephalopathy
* Females who are breastfeeding
* Positive serum pregnancy test at any time during the study (female of childbearing potential)
* Participants receiving ongoing therapy with any disallowed medication
* Current alcohol or substance use judged by the investigator to potentially interfere with study compliance
* Malignancy other than cutaneous Kaposi's sarcoma or basal cell carcinoma
* Active, serious infections (other than HIV-1 infection) requiring parenteral antibiotic or antifungal therapy within 30 days prior to baseline
* Participation in any other clinical trial (except for the etravirine or maraviroc expanded access program), without prior approval from sponsor
* Any other clinical condition or prior therapy that would make participants unsuitable for the study
* Known hypersensitivity to study drug, metabolites or formulation excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 724 (Actual)
Dates: Start 2008-07; Primary Completion 2010-12 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Szwarcberg, MD, MPH, Study Director — Gilead Sciences
Locations (180):
- United States (94):
  - Southwest Center for HIV/AIDS, Phoenix, Arizona
  - Health for Life Clinic, PLLC, Little Rock, Arkansas
  - Pacific Oaks Medical Group, Beverly Hills, California
  - AIDS Healthcare Foundation-Research Center, Beverly Hills, California
  - Center for Special Immunology, Fountain Valley, California
  - The Living Hope Foundation, Long Beach, California
  - Kaiser Permanente, Los Angeles, California
  - Jeffrey Goodman Special Care Clinic, Los Angeles, California
  - University of Southern California, AIDS Clinical Trials Unit, Los Angeles, California
  - Peter J. Ruane, MD, Inc., Los Angeles, California
  - Tony Mills, MD Internal Medicine, Los Angeles, California
  - Orange Coast Medical Group, Newport Beach, California
  - Alameda County Medical Center, Oakland, California
  - East Bay AIDS Center, Oakland, California
  - Kaiser Permanente, Sacramento, California
  - David J. Shamblaw, MD Inc., San Diego, California
  - Metropolis Medical, San Francisco, California
  - San Francisco VA Medical Center/UCSF, San Francisco, California
  - Connecticut Health Care Group, Glastonbury, Connecticut
  - Circle Medical LLC, Norwalk, Connecticut
  - The Stamford Hospital - Stamford ID, Stamford, Connecticut
  - Whitman-Walker Clinic, Washington D.C., District of Columbia
  - The George Washington University Medical Center, Washington D.C., District of Columbia
  - South Florida Clinical Research, Atlantis, Florida
  - Lifeway , Inc., Fort Lauderdale, Florida
  - NorthPoint Medical, Fort Lauderdale, Florida
  - Therafirst Medical Centers, Fort Lauderdale, Florida
  - Broward Health CCC, Fort Lauderdale, Florida
  - Gary Richmond, MD, PA, Inc., Fort Lauderdale, Florida
  - Associates In Infectious Diseases, Ft. Pierce, Florida
  - The Kinder Medical Group, Miami, Florida
  - University of Miami, Miami, Florida
  - Wohlfeiler, Piperato and Associates, LLC, North Miami Beach, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Infectious Disease of Central Florida, Orlando, Florida
  - Barry M. Rodwick, M. D., Safety Harbor, Florida
  - St. Joseph's Comprehensive Research Institute, Tampa, Florida
  - Treasure Coast Infectious Disease Consultants, Vero Beach, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - The Emory Clinic, Inc., Division of Infectious Diseases, Atlanta, Georgia
  - Atlanta ID Group, Atlanta, Georgia
  - Infectious Disease Specialists of Atlanta (IDSA), Decatur, Georgia
  - Mercer Univ. School of Medicine, Macon, Georgia
  - Chatham County Health Department, Savannah, Georgia
  - Hawaii AIDS Clinical Research Program HACRP, Honolulu, Hawaii
  - The Ruth M. Rothstein CORE Center, Chicago, Illinois
  - Howard Brown Health Center, Chicago, Illinois
  - Northstar Medical Center, Chicago, Illinois
  - University of Kentucky Healthcare/Bluegrass Care Clinic, Lexington, Kentucky
  - University of Maryland, Institute of Human Virology, Baltimore, Maryland
  - Community Research Initiative of New England, Boston, Massachusetts
  - Be Well Medical Center, Berkley, Michigan
  - Wayne State University, Detroit, Michigan
  - Henry Ford Hospital Div of Infectious Disease, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Southampton Healthcare, Inc., St Louis, Missouri
  - ID Care, Hillsborough, New Jersey
  - Saint Michael's Medical Center, Newark, New Jersey
  - University of Medicine and Dentistry of New Jersey; University Hospital Infectious Disease Practice, Newark, New Jersey
  - South Jersey Infectious Disease, Somer Point, New Jersey
  - Southwest C.A.R.E. Center, Santa Fe, New Mexico
  - Albany Medical College, Albany, New York
  - STAR Health Care Center, Brooklyn, New York
  - Greiger Clinic, Mount Vernon, New York
  - Beth Israel Medical Center, New York, New York
  - Chelsea Village Medical, PC, New York, New York
  - Ricky K. Hsu, MD, PC, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - AIDS Community HealthCenter, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina/ School of Medicine Division of Infectious Diseases/ AIDS Clinical Trials Unit, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Brody School of Medicine at East Carolina University, Greenville, North Carolina
  - Rosedale Infectious Diseases, Huntersville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Summa Health CARE Center, Akron, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - Thomas Jefferson University Jefferson Alumni Hall, Philadelphia, Pennsylvania
  - Central Texas Clinical Research, Austin, Texas
  - AIDS Arms/ Peabody Health Center, Dallas, Texas
  - Southwest Infectious Disease Clinical Research, Dallas, Texas
  - Presbyterian Hospital of Dallas, Dallas, Texas
  - North Texas Infectious Disease Consultants, Dallas, Texas
  - Tarrant County Infectious Disease Associates, Fort Worth, Texas
  - Garcia Family Health Group, Harlingen, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Gordon E. Crofoot, MD, PA, Houston, Texas
  - The Schrader Clinic, Houston, Texas
  - Joseph C. Gathe, JR. MD, F.A.C.P., Houston, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - Clinical Alliance for Research & Education - Infectious Diseases, LLC (CARE-ID), Annandale, Virginia
  - EHS Pulmonary and Critical Care, Spokane, Washington
- Australia (8):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Ground Zero Medical Centre, Darlinghurst, New South Wales
  - Holdsworth House Medical Practice, Darlinghurst, New South Wales
  - St. Vincent's Hospital, Sydney, Darlinghurst, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Albion Street Centre, Sydney, New South Wales
  - East Sidney Doctors, Sydney, New South Wales
  - Westmead Hospital, Wentworthville, New South Wales
- Belgium (5):
  - Institute of Tropical Medicine, Antwerp
  - C.H.U. St Pierre, Brussels
  - Hôpital Erasme, Brussels
  - CHU de Charleroi-Hopital civil, Charleroi
  - Centre Hospitalier Universitaire de Liège, Liège
- Canada (9):
  - Downtown Infectious Diseases Clinic, Vancouver, British Columbia
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - CascAids Research, Toronto, Ontario
  - Canadian Immunodeficiency Research Collaborative (CIRC) Inc., Toronto, Ontario
  - University Health Network, Toronto General Hospital, Toronto, Ontario
  - Clinique medicale l'Actuel, Montreal, Quebec
  - Immunodeficiency Service, McGill University Health Centre (MUHC), Montreal, Quebec
  - University of Manitoba - Health Sciences Centre, Winnipeg
- France (11):
  - Hopital de Bicentre - Service de medecine Interne et Immunologie, Le Kremlin-Bicêtre
  - University Hospital of Montpellier - Gui de Chauliac, Montpellier
  - CHU Nantes, Nantes
  - C.H.U. de Nice - Hopital de l'Archet 1, Nice
  - Hopital Saint Louis, Paris
  - Hopital Saint Antoine - Infectious Desease Department, Paris
  - Hopital Pitie Salpetriere - Infectious Deseases Department, Paris
  - APHP Hopital Bichat-Claude Bernard, Paris
  - Hopital Tenon, Paris
  - CHU Bordeaux, Pessac
  - Hopital Purpan - Service of Infectious Diseases, Toulouse
- Germany (9):
  - Universitatsklinikum Bonn, Bonn
  - Klinikum der Universitat zu Koln, Cologne
  - Universitatsklinikum Dusseldorf, Düsseldorf
  - Universitatklinikum Essen, Essen
  - Klinikum der J.W. Goethe-Universitat, Frankfurt
  - IFI-Institute, Hamburg
  - Ambulanzzentrum am Universitatsklinikum Hamburg Eppendorf, Hamburg
  - Medizinische Universitatsklinik Kiel, Kiel
  - MUC Research, Munich
- Italy (8):
  - Ospedali Riuniti Di Bergamo, Bergamo
  - Spedali Civili di Brescia, Brescia
  - Fondazione Centro San Raffaele del Monte Tabor, Milan
  - Ospedale L. Sacco, Milan
  - Ospedale Luigi Sacco, Milan
  - Istituto Nazionale per le Malattie Infettive Lazzaro Spallanzani I.R.C.C.S., Rome
  - Universita La Sapienza Policlinico Umberto I, Rome
  - Universita' Cattolica Del Sacro Cuore, Rome
- Mexico (4):
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (INCMYNSZ), México, D.f.
  - Hospital Regional de Leon Guanajuato, León, Guanajuato
  - Hospital Civil de Guadalajara, Guadalajara, Jalisco
  - Hospital Central Morones Prieto, San Luis Potosí City, San Luis Potsi
- Erasmus Medisch Centrum, Rotterdam, Netherlands
- Portugal (5):
  - Hospital Fernando Fonseca, Amadora
  - Hospital Santo Antonio dos Capuchos, Lisbon
  - Hospital de Santa Maria, Lisbon
  - Hospital Pulido Valente, Lisbon
  - Hospital de Sao Joao, Porto
- Puerto Rico (5):
  - Instituto de Investigacion Cientifica del Sur, Ponce
  - Clinical Research Puerto Rico, Inc., San Juan
  - HOPE Clinical Research, San Juan
  - VA Caribbean healthcare System, San Juan
  - University of Puerto Rico, School of Medicine, Proyecto ACTU, San Juan
- Spain (16):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Universitario Germans Trias i Pujol, Barcelona
  - Hospital Reina Sofia, Córdoba
  - Hospital General Universitario del Elche, Elche
  - Hospital Clinico San Cecilio, Granada
  - Hospital La Princesa, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Doce De Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Virgen del Rocio, Seville
  - Complexo Hospitalario Xeral-Cies (Chuvi) Vigo, Vigo
- Universitatsspital Zurich, Zurich, Switzerland
- United Kingdom (4):
  - RIDU, Western General Hospital, Edinburgh
  - Imperial College Healthcare NHS Trust, St. Mary's Campus, London
  - Royal Free and University College Medical School, London
  - North Manchester General Hospital, Manchester

REFERENCES:
- [Result] Molina JM, Lamarca A, Andrade-Villanueva J, Clotet B, Clumeck N, Liu YP, Zhong L, Margot N, Cheng AK, Chuck SL; Study 145 Team. Efficacy and safety of once daily elvitegravir versus twice daily raltegravir in treatment-experienced patients with HIV-1 receiving a ritonavir-boosted protease inhibitor: randomised, double-blind, phase 3, non-inferiority study. Lancet Infect Dis. 2012 Jan;12(1):27-35. doi: 10.1016/S1473-3099(11)70249-3. Epub 2011 Oct 18. PMID 22015077

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in a total of 161 study sites in Australia, Europe, and North America. The first participant was screened on 19 June 2008. The last study visit occurred on 22 April 2015.
Pre-assignment Details: 1335 participants were screened.
Groups:
- Elvitegravir: Elvitegravir (EVG) 85 or 150 mg tablet once daily plus raltegravir (RAL) placebo plus background regimen (1 fully-active ritonavir (RTV)-boosted protease inhibitor (PI) plus 1 or 2 additional agents) in the Randomized Phase, followed by EVG 85 or 150 mg tablet once daily plus background regimen in the Open-Label Phase.
- Raltegravir: RAL 400 mg tablet twice daily plus EVG placebo plus background regimen (1 fully-active RTV-boosted PI plus 1 or 2 additional agents) in the Randomized Phase, followed by EVG 85 or 150 mg tablet once daily plus background regimen in the Open-Label Phase.
Period: Randomized Phase
Arm/Group | Elvitegravir | Raltegravir
Started | 361 | 363
Randomized and Treated | 354 | 358
Completed | 205 | 209
Not Completed | 156 | 154
Not completed — Randomized but Not Treated | 7 | 5
Not completed — Participant Noncompliance | 40 | 32
Not completed — Lost to Follow-up | 34 | 34
Not completed — Withdrew Consent | 31 | 22
Not completed — Lack of Efficacy | 14 | 19
Not completed — Protocol Violation | 10 | 11
Not completed — Adverse Event | 8 | 12
Not completed — Investigator's Discretion | 7 | 10
Not completed — Death | 2 | 9
Not completed — Pregnancy | 3 | 0
Period: Open-Label Phase
Arm/Group | Elvitegravir | Raltegravir
Started | 196 (9 participants completing the Randomized Phase did not continue to the Open-Label Phase.) | 151 (58 participants completing the Randomized Phase did not continue to the Open-Label Phase.)
Completed | 152 | 121
Not Completed | 44 | 30
Not completed — Lost to Follow-up | 10 | 8
Not completed — Withdrew Consent | 12 | 6
Not completed — Participant Noncompliance | 7 | 7
Not completed — Lack of Efficacy | 7 | 4
Not completed — Investigator's Discretion | 3 | 2
Not completed — Death | 3 | 1
Not completed — Adverse Event | 1 | 2
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were randomized and received at least one dose of study drug
Groups:
- Elvitegravir: EVG 85 or 150 mg tablet once daily plus RAL placebo plus background regimen (1 fully-active RTV-boosted PI plus 1 or 2 additional agents) in the Randomized Phase, followed by EVG 85 or 150 mg tablet once daily plus background regimen in the Open-Label Phase.
- Total: Total of all reporting groups
Arm/Group | Elvitegravir | Raltegravir | Total
Number analyzed (Participants) | 354 | 358 | 712
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (9.0) | 45 (9.1) | 45 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 67 | 127
  Male | 294 | 291 | 585
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 81 | 74 | 155
  Not Hispanic or Latino | 272 | 283 | 555
  Unknown or Not Reported | 1 | 1 | 2
Race/Ethnicity, Customized [Number; unit: participants]
  White | 210 | 227 | 437
  Black or African American | 128 | 119 | 247
  Asian | 9 | 5 | 14
  American Indian or Alaska Native | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Other | 3 | 4 | 7
Region of Enrollment [Number; unit: participants] — All randomized participants were analyzed for Region of Enrollment (elvitegravir arm: n = 361; raltegravir arm: n = 363)
  participants
    United States | 230 | 223 | 453
    Portugal | 10 | 11 | 21
    Spain | 14 | 20 | 34
    United Kingdom | 6 | 5 | 11
    Italy | 7 | 10 | 17
    France | 16 | 9 | 25
    Mexico | 26 | 25 | 51
    Canada | 16 | 18 | 34
    Puerto Rico | 8 | 14 | 22
    Belgium | 5 | 6 | 11
    Australia | 17 | 12 | 29
    Germany | 6 | 8 | 14
    Netherlands | 0 | 2 | 2
HIV-1 RNA [Mean (Standard Deviation); unit: log10 copies/mL] | 4.26 (0.969) | 4.27 (0.943) | 4.26 (0.955)
HIV-1 RNA category [Number; unit: participants]
  ≤ 100,000 copies/mL | 263 | 267 | 530
  > 100,000 copies/mL | 91 | 91 | 182
Cluster of differentiation (CD4) Cell Count [Mean (Standard Deviation); unit: cells/mm^3] | 257.9 (204.31) | 265.3 (207.04) | 261.6 (205.57)
HIV Disease Status [Number; unit: participants]
  Asymptomatic | 172 | 175 | 347
  Symptomatic HIV Infections | 52 | 54 | 106
  AIDS | 126 | 125 | 251
  Unknown | 4 | 4 | 8
Type of PI in Background Regimen (Excluding Ritonavir) [Number; unit: participants] — One participant in the Raltegravir group switched from darunavir to fosamprenavir at Day 5, and is counted only in the number receiving darunavir at baseline.
  participants
    atazanavir | 64 | 53 | 117
    darunavir | 202 | 206 | 408
    fosamprenavir | 14 | 20 | 34
    lopinavir | 68 | 72 | 140
    tipranavir | 6 | 7 | 13
Type of NRTI in Background Regimen [Number; unit: participants]
  tenofovir disoproxil fumarate | 163 | 171 | 334
  emtricitabine/tenofovir disoproxil fumarate | 91 | 66 | 157
  lamivudine | 13 | 13 | 26
  abacavir | 6 | 15 | 21
  abacavir/lamivudine | 4 | 8 | 12
  lamivudine/zidovudine | 6 | 5 | 11
  zidovudine | 3 | 6 | 9
  didanosine | 1 | 7 | 8
  emtricitabine | 2 | 3 | 5
  no NRTI in background regimen | 65 | 64 | 129
Enfuvirtide (T-20) in background regimen [Number; unit: participants]
  No | 352 | 357 | 709
  Yes | 2 | 1 | 3
Etravirine in background regimen [Number; unit: participants]
  No | 309 | 303 | 612
  Yes | 45 | 55 | 100
Maraviroc in background regimen [Number; unit: participants]
  No | 330 | 340 | 670
  Yes | 24 | 18 | 42
Phenotypic Sensitivity Score [Number; unit: participants] — Phenotypic sensitivity score (PSS) was calculated by summing up drug susceptibility values (1=sensitive; 0.5=partially sensitive; 0=resistance or reduced susceptibility) on all drugs in the baseline background regimen. For subjects naive to enfuvirtide (or maraviroc), a score of 1 was assigned for enfuvirtide (or maraviroc). Higher scores correspond to increased sensitivity.
  participants
    1.0 | 5 | 4 | 9
    1.5 | 23 | 28 | 51
    2.0 | 309 | 313 | 622
    2.5 | 2 | 1 | 3
    3.0 | 14 | 10 | 24
    3.5 | 0 | 1 | 1
    No baseline PSS score | 1 | 1 | 2
Chronic Hepatitis B (HBV) Infection Status [Number; unit: participants]
  Indeterminant | 1 | 0 | 1
  Negative | 333 | 342 | 675
  Positive | 17 | 13 | 30
  No baseline HBV measurement | 3 | 3 | 6
Chronic Hepatitis C (HCV) Infection Status [Number; unit: participants]
  Indeterminant | 2 | 2 | 4
  Negative | 305 | 298 | 603
  Positive | 44 | 55 | 99
  No baseline HCV measurement | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving and Maintaining Confirmed HIV-1 RNA < 50 Copies/mL at Week 48
Description: The percentage of participants achieving and maintaining confirmed HIV-1 RNA < 50 copies/mL at Week 48 was analyzed using the FDA-defined Time to Loss of Virologic Response (TLOVR) algorithm, which takes into account a patient's longitudinal viral load up to the predefined time point by considering patterns of suppression and rebounding.
Time Frame: Week 48
Population: ITT Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Elvitegravir | Raltegravir
Number analyzed (Participants) | 351 | 351
percentage of participants | 59.0 | 57.8
Statistical Analysis 1: Comparison: Elvitegravir vs Raltegravir; The planned sample size of 700 HIV-1 infected participants, (350 in each group) was estimated to provide at least 85% power to establish noninferiority in the percentage of participants achieving and maintaining confirmed HIV-1 RNA < 50 copies/mL through Week 48. For sample size and power computation, it was assumed that both elvitegravir and raltegravir arms have a response rate of 0.74, that a noninferiority margin was 0.10, and that the significance level of the test was 1-sided 0.025 level; Test type: Non-Inferiority or Equivalence — Null hypothesis: the EVG group was at least 10% worse than the RAL group with respect to percentage of participants achieving and maintaining HIV-1 RNA < 50 copies/mL through Week 48; alternative hypothesis: the EVG group was less than 10% worse than the RAL group; Difference in percentages = 1.1, 95% CI 2-sided [-6.0 to 8.2] — The difference in percentages and its 95% confidence interval (CI) were based on stratum-adjusted HIV-1 RNA level and the class of second agent (NRTI or other classes) using Mantel-Haenszel (MH) proportions and normal approximation

2. Secondary Outcome: Percentage of Participants Achieving and Maintaining Confirmed HIV-1 RNA < 50 Copies/mL at Week 96
Description: The percentage of participants achieving and maintaining confirmed HIV-1 RNA < 50 copies/mL at Week 96 was analyzed using the FDA-defined TLOVR algorithm, which takes into account a patient's longitudinal viral load up to the predefined time point by considering patterns of suppression and rebounding.
Time Frame: Week 96
Population: ITT Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Elvitegravir | Raltegravir
Number analyzed (Participants) | 351 | 351
percentage of participants | 47.6 | 45.0
Statistical Analysis 1: Comparison: Elvitegravir vs Raltegravir; Test type: Non-Inferiority or Equivalence — Null hypothesis: the EVG arm was at least 10% worse than the RAL arm with respect to percentage of participants achieving and maintaining HIV-1 RNA < 50 copies/mL through Week 48; alternative hypothesis: the EVG arm was less than 10% worse than the RAL arm; Difference in percentages = 2.6, 95% CI 2-sided [-4.6 to 9.9] — The difference in percentages and its 95% CI were based on stratum-adjusted HIV-1 RNA level and the class of second agent (NRTI or other classes) using MH proportions and normal approximation

3. Secondary Outcome: Percentage of Participants Achieving and Maintaining Confirmed HIV-1 RNA < 400 Copies/mL at Week 48
Description: The percentage of participants achieving and maintaining confirmed HIV-1 RNA < 400 copies/mL at Week 48 was analyzed using the FDA-defined TLOVR algorithm, which takes into account a patient's longitudinal viral load up to the predefined time point by considering patterns of suppression and rebounding.
Time Frame: Week 48
Population: ITT Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Elvitegravir | Raltegravir
Number analyzed (Participants) | 351 | 351
percentage of participants | 68.1 | 67.2
Statistical Analysis 1: Comparison: Elvitegravir vs Raltegravir; Test type: Superiority or Other; Difference in percentages = 0.9, 95% CI 2-sided [-6.0 to 7.7] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Percentage of Participants Achieving and Maintaining Confirmed HIV-1 RNA < 400 Copies/mL at Week 96
Description: The percentage of participants achieving and maintaining confirmed HIV-1 RNA < 400 copies/mL at Week 96 was analyzed using the FDA-defined TLOVR algorithm, which takes into account a patient's longitudinal viral load up to the predefined time point by considering patterns of suppression and rebounding.
Time Frame: Week 96
Population: ITT Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Elvitegravir | Raltegravir
Number analyzed (Participants) | 351 | 351
percentage of participants | 57.0 | 56.1
Statistical Analysis 1: Comparison: Elvitegravir vs Raltegravir; Test type: Superiority or Other; Difference in percentages = 0.9, 95% CI 2-sided [-6.4 to 8.2] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Virologic Response at Week 48 (HIV-1 RNA < 50 Copies/mL)
Description: Virologic response at Week 48 (percentage of participants with HIV-1 RNA < 50 copies/mL) was analyzed using the FDA-defined Snapshot algorithm, which defines a patient's virologic response status using the viral load along with study drug discontinuation status at the predefined time point within an allowed window of time.
Time Frame: Week 48
Population: ITT Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Elvitegravir | Raltegravir
Number analyzed (Participants) | 351 | 351
percentage of participants | 59.8 | 57.5
Statistical Analysis 1: Comparison: Elvitegravir vs Raltegravir; Test type: Superiority or Other; Difference in percentages = 2.2, 95% CI 2-sided [-5.0 to 9.3] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Virologic Response at Week 96 (HIV-1 RNA < 50 Copies/mL)
Description: Virologic response at Week 96 (percentage of participants with HIV-1 RNA < 50 copies/mL) was analyzed using the FDA-defined Snapshot algorithm, which defines a patient's virologic response status using the viral load along with study drug discontinuation status at the predefined time point within an allowed window of time.
Time Frame: Week 96
Population: ITT Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Elvitegravir | Raltegravir
Number analyzed (Participants) | 351 | 351
percentage of participants | 52.4 | 53.0
Statistical Analysis 1: Comparison: Elvitegravir vs Raltegravir; Test type: Superiority or Other; Difference in percentages = -0.5, 95% CI 2-sided [-7.9 to 6.8] — [estimate comment as in outcome 2, analysis 1]

7. Secondary Outcome: Percentage of Participants With Pure Virologic Failure (HIV-1 RNA Cutoff at 50 Copies/mL) up to Week 48
Description: The percentage of participants with pure virologic failure (HIV-1 RNA cutoff at 50 copies/mL) up to Week 48 was estimated using the Kaplan-Meier method in the time to event analysis.
Time Frame: Baseline to Week 48
Population: ITT Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Elvitegravir | Raltegravir
Number analyzed (Participants) | 351 | 351
percentage of participants | 35 [29.8 to 39.8] | 35 [29.8 to 39.8]

8. Secondary Outcome: Percentage of Participants With Pure Virologic Failure (HIV-1 RNA Cutoff at 50 Copies/mL) up to Week 96
Description: The percentage of participants with pure virologic failure (HIV-1 RNA cutoff at 50 copies/mL) up to Week 96 was estimated using the Kaplan-Meier method in the time to event analysis.
Time Frame: Baseline to Week 96
Population: ITT Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Elvitegravir | Raltegravir
Number analyzed (Participants) | 351 | 351
percentage of participants | 45 [39.3 to 49.9] | 46 [41.1 to 51.9]

9. Secondary Outcome: Percentage of Participants With Pure Virologic Failure (HIV-1 RNA Cutoff at 400 Copies/mL) up to Week 48
Description: The percentage of participants with pure virologic failure (HIV-1 RNA cutoff at 400 copies/mL) up to Week 48 was estimated using the Kaplan-Meier method in the time to event analysis.
Time Frame: Baseline to Week 48
Population: ITT Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Elvitegravir | Raltegravir
Number analyzed (Participants) | 351 | 351
percentage of participants | 24 [19.5 to 28.5] | 24 [19.7 to 28.9]

10. Secondary Outcome: Percentage of Participants With Pure Virologic Failure (HIV-1 RNA Cutoff at 400 Copies/mL) up to Week 96
Description: The percentage of participants with pure virologic failure (HIV-1 RNA cutoff at 400 copies/mL) up to Week 96 was estimated using the Kaplan-Meier method in the time to event analysis.
Time Frame: Baseline to Week 96
Population: ITT Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Elvitegravir | Raltegravir
Number analyzed (Participants) | 351 | 351
percentage of participants | 32 [26.7 to 36.7] | 31 [26.1 to 36.1]

11. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 48
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 48 was analyzed using the missing = failure method, where participants with missing data were considered as having failed to meet the criteria for evaluation.
Time Frame: Week 48
Population: ITT Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Elvitegravir | Raltegravir
Number analyzed (Participants) | 351 | 351
percentage of participants | 61.0 | 60.7
Statistical Analysis 1: Comparison: Elvitegravir vs Raltegravir; Test type: Superiority or Other; Difference in percentages = 0.2, 95% CI 2-sided [-6.9 to 7.3] — [estimate comment as in outcome 2, analysis 1]

12. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 96
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 96 was analyzed using the missing = failure method.
Time Frame: Week 96
Population: ITT Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Elvitegravir | Raltegravir
Number analyzed (Participants) | 351 | 351
percentage of participants | 53.6 | 56.4
Statistical Analysis 1: Comparison: Elvitegravir vs Raltegravir; Test type: Superiority or Other; Difference in percentages = -2.9, 95% CI 2-sided [-10.2 to 4.4] — [estimate comment as in outcome 2, analysis 1]

13. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 400 Copies/mL at Week 48
Description: The percentage of participants with HIV-1 RNA < 400 copies/mL at Week 48 was analyzed using the missing = failure method.
Time Frame: Week 48
Population: ITT Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Elvitegravir | Raltegravir
Number analyzed (Participants) | 351 | 351
percentage of participants | 70.1 | 72.1
Statistical Analysis 1: Comparison: Elvitegravir vs Raltegravir; Test type: Superiority or Other; Difference in percentages = -2.0, 95% CI 2-sided [-8.6 to 4.7] — [estimate comment as in outcome 2, analysis 1]

14. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 400 Copies/mL at Week 96
Description: The percentage of participants with HIV-1 RNA < 400 copies/mL at Week 96 was analyzed using the missing = failure method.
Time Frame: Week 96
Population: ITT Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Elvitegravir | Raltegravir
Number analyzed (Participants) | 351 | 351
percentage of participants | 61.3 | 63.0
Statistical Analysis 1: Comparison: Elvitegravir vs Raltegravir; Test type: Superiority or Other; Difference in percentages = -1.7, 95% CI 2-sided [-8.8 to 5.5] — [estimate comment as in outcome 2, analysis 1]

15. Secondary Outcome: Change From Baseline in HIV-1 RNA at Week 48
Description: The change from baseline in log10 HIV-1 RNA (copies/mL) at Week 48 was analyzed.
Time Frame: Baseline to Week 48
Population: Participants in the ITT Analysis Set with evaluable change data at Week 48 were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Elvitegravir | Raltegravir
Number analyzed (Participants) | 280 | 291
log10 copies/mL | -2.17 (1.162) | -2.18 (1.178)
Statistical Analysis 1: Comparison: Elvitegravir vs Raltegravir; Test type: Superiority or Other; Difference in log10 copies/mL = 0.01, 95% CI 2-sided [-0.16 to 0.19] — The difference in least squares means (LSM) and its 95% CI were obtained using an analysis of variance model (ANOVA) adjusting for baseline HIV-1 RNA level and class of the second agent (NRTI or other classes)

16. Secondary Outcome: Change From Baseline in HIV-1 RNA at Week 96
Description: The change from baseline in log10 HIV-1 RNA (copies/mL) at Week 96 was analyzed.
Time Frame: Baseline to Week 96
Population: Participants in the ITT Analysis Set with evaluable change data at Week 96 were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Elvitegravir | Raltegravir
Number analyzed (Participants) | 238 | 238
log10 copies/mL | -2.26 (1.078) | -2.31 (1.068)
Statistical Analysis 1: Comparison: Elvitegravir vs Raltegravir; Test type: Superiority or Other; Difference in log10 copies/mL = 0.05, 95% CI 2-sided [-0.12 to 0.22] — The difference in LSM and its 95% CI were obtained using ANOVA adjusting for baseline HIV-1 RNA level and class of the second agent (NRTI or other classes)

17. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 48
Description: The change from baseline in CD4 cell count (cells/mm^3) at Week 48 was analyzed.
Time Frame: Baseline to Week 48
Population: Participants in the ITT Analysis Set with evaluable change data at Week 48 were analyzed.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Elvitegravir | Raltegravir
Number analyzed (Participants) | 267 | 282
cells/mm^3 | 138 (141.4) | 147 (148.9)
Statistical Analysis 1: Comparison: Elvitegravir vs Raltegravir; Test type: Superiority or Other; Difference in cells/mm^3 = -9, 95% CI 2-sided [-33 to 16] — [estimate comment as in outcome 16, analysis 1]

18. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 96
Description: The change from baseline in CD4 cell count (cells/mm^3) at Week 96 was analyzed.
Time Frame: Baseline to Week 96
Population: Participants in the ITT Analysis Set with evaluable change data at Week 96 were analyzed.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Elvitegravir | Raltegravir
Number analyzed (Participants) | 231 | 233
cells/mm^3 | 205 (191.5) | 198 (162.2)
Statistical Analysis 1: Comparison: Elvitegravir vs Raltegravir; Test type: Superiority or Other; Difference in cells/mm^3 = 7, 95% CI 2-sided [-25 to 39] — [estimate comment as in outcome 16, analysis 1]

ADVERSE EVENTS:
Time Frame: Baseline through end of study drug treatment (average exposure: 100 weeks) plus 30 days
Description: Safety Analysis Set: participants who were randomized and received at least one dose of study drug
Groups:
- Elvitegravir: Adverse events in this reporting group are those experienced by participants in the Elvitegravir group during the Randomized Phase
  EVG 85 or 150 mg tablet once daily plus RAL placebo plus background regimen (1 fully-active RTV-boosted PI plus 1 or 2 additional agents) in the Randomized Phase, followed by EVG 85 or 150 mg tablet once daily plus background regimen in the Open-Label Phase.
- Raltegravir: Adverse events in this reporting group are those experienced by participants in the Raltegravir group during the Randomized Phase
  RAL 400 mg tablet twice daily plus EVG placebo plus background regimen (1 fully-active RTV-boosted PI plus 1 or 2 additional agents) in the Randomized Phase, followed by EVG 85 or 150 mg tablet once daily plus background regimen in the Open-Label Phase.
- All Elvitegravir: Adverse events in this reporting group are those experienced by participants in the Elvitegravir group during both the Randomized Phase and Open-Label Phase, and those experienced by participants in the Raltegravir group following switch to EVG in the Open-Label Phase only.
Arm/Group | Elvitegravir | Raltegravir | All Elvitegravir
Serious Adverse Events (participants affected / at risk) | 73/354 | 86/358 | 127/505
Other Adverse Events (participants affected / at risk) | 279/354 | 250/358 | 394/505
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Elvitegravir (N=354) | Raltegravir (N=358) | All Elvitegravir (N=505)
Coombs positive haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 0 | 3
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 2
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 1
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 2 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1
Mitral valve prolapse (Cardiac disorders) | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 2 | 3
Pericardial effusion (Cardiac disorders) | 1 | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Haemophilia (Congenital, familial and genetic disorders) | 0 | 1 | 0
Phimosis (Congenital, familial and genetic disorders) | 1 | 0 | 1
Basedow's disease (Endocrine disorders) | 0 | 0 | 1
Cushing's syndrome (Endocrine disorders) | 0 | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 1
Anogenital dysplasia (Gastrointestinal disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 1 | 2
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1
Chest pain (General disorders) | 1 | 4 | 4
Drug withdrawal syndrome (General disorders) | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Chronic hepatic failure (Hepatobiliary disorders) | 1 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 2 | 0
Hepatitis cholestatic (Hepatobiliary disorders) | 1 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Immune reconstitution inflammatory syndrome (Immune system disorders) | 1 | 0 | 1
Abscess limb (Infections and infestations) | 1 | 0 | 1
Acute hepatitis B (Infections and infestations) | 0 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
Arthritis infective (Infections and infestations) | 0 | 1 | 0
Biliary sepsis (Infections and infestations) | 0 | 1 | 0
Breast abscess (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 2 | 4 | 3
Bursitis infective (Infections and infestations) | 0 | 0 | 1
Candida infection (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 5 | 5 | 8
Enterocolitis bacterial (Infections and infestations) | 0 | 0 | 1
Epididymitis (Infections and infestations) | 1 | 0 | 1
Extradural abscess (Infections and infestations) | 1 | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 3
Genital herpes (Infections and infestations) | 0 | 1 | 1
Hepatitis A (Infections and infestations) | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 1
Infectious colitis (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1
Liver abscess (Infections and infestations) | 0 | 0 | 1
Meningitis aseptic (Infections and infestations) | 1 | 0 | 1
Muscle abscess (Infections and infestations) | 0 | 1 | 0
Neurosyphilis (Infections and infestations) | 1 | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 1 | 0 | 1
Ophthalmic herpes zoster (Infections and infestations) | 1 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 1
Parotid abscess (Infections and infestations) | 0 | 1 | 0
Periorbital cellulitis (Infections and infestations) | 1 | 0 | 1
Perirectal abscess (Infections and infestations) | 0 | 0 | 1
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 12 | 7 | 15
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 2
Postoperative wound infection (Infections and infestations) | 1 | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0 | 3
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 1 | 0 | 2
Skin infection (Infections and infestations) | 1 | 0 | 1
Spinal cord abscess (Infections and infestations) | 0 | 1 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 3
Urosepsis (Infections and infestations) | 1 | 1 | 1
Viral infection (Infections and infestations) | 1 | 0 | 2
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 2
Chemical poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Foreign body (Injury, poisoning and procedural complications) | 0 | 0 | 1
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 2 | 2 | 3
Perirenal haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 2 | 0
Skull fractured base (Injury, poisoning and procedural complications) | 0 | 0 | 1
Splenic injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 2
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 2
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 3
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperosmolar hyperglycaemic state (Metabolism and nutrition disorders) | 0 | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Anal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Anal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hodgkin's disease stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Oral papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Primary effusion lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Queyrat erythroplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1 | 0
Carotid artery dissection (Nervous system disorders) | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 2 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 1
Embolic stroke (Nervous system disorders) | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 1 | 1 | 1
Hemiparesis (Nervous system disorders) | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
Partial seizures (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 1 | 2 | 3
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 3
Syncope (Nervous system disorders) | 2 | 0 | 7
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 1
Unresponsive to stimuli (Nervous system disorders) | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Acute psychosis (Psychiatric disorders) | 0 | 0 | 1
Alcohol abuse (Psychiatric disorders) | 0 | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 1
Drug dependence (Psychiatric disorders) | 1 | 0 | 1
Hallucination, auditory (Psychiatric disorders) | 1 | 0 | 1
Homicidal ideation (Psychiatric disorders) | 1 | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0
Substance abuse (Psychiatric disorders) | 1 | 1 | 1
Suicidal ideation (Psychiatric disorders) | 3 | 4 | 4
Suicide attempt (Psychiatric disorders) | 1 | 1 | 2
Acute kidney injury (Renal and urinary disorders) | 2 | 1 | 5
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 2 | 0
Obstructive uropathy (Renal and urinary disorders) | 0 | 0 | 1
Renal tubular acidosis (Renal and urinary disorders) | 1 | 0 | 1
Renal vein thrombosis (Renal and urinary disorders) | 1 | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Aortic stenosis (Vascular disorders) | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 1
Haemodynamic instability (Vascular disorders) | 1 | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 1
Peripheral artery thrombosis (Vascular disorders) | 1 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0
Shock (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Elvitegravir (N=354) | Raltegravir (N=358) | All Elvitegravir (N=505)
Abdominal pain (Gastrointestinal disorders) | 24 | 18 | 40
Diarrhoea (Gastrointestinal disorders) | 120 | 77 | 158
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 14 | 9 | 28
Nausea (Gastrointestinal disorders) | 45 | 41 | 61
Vomiting (Gastrointestinal disorders) | 22 | 28 | 30
Fatigue (General disorders) | 39 | 25 | 55
Pyrexia (General disorders) | 18 | 19 | 29
Bronchitis (Infections and infestations) | 34 | 34 | 57
Folliculitis (Infections and infestations) | 18 | 7 | 25
Gastroenteritis (Infections and infestations) | 15 | 7 | 28
Influenza (Infections and infestations) | 15 | 10 | 30
Nasopharyngitis (Infections and infestations) | 40 | 32 | 56
Oral herpes (Infections and infestations) | 15 | 6 | 26
Sinusitis (Infections and infestations) | 28 | 28 | 48
Upper respiratory tract infection (Infections and infestations) | 75 | 59 | 116
Urinary tract infection (Infections and infestations) | 28 | 35 | 52
Hypercholesterolaemia (Metabolism and nutrition disorders) | 12 | 20 | 26
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 | 28 | 57
Back pain (Musculoskeletal and connective tissue disorders) | 42 | 36 | 68
Muscle spasms (Musculoskeletal and connective tissue disorders) | 18 | 13 | 28
Myalgia (Musculoskeletal and connective tissue disorders) | 14 | 11 | 26
Pain in extremity (Musculoskeletal and connective tissue disorders) | 28 | 25 | 48
Headache (Nervous system disorders) | 49 | 37 | 63
Anxiety (Psychiatric disorders) | 16 | 9 | 33
Depression (Psychiatric disorders) | 33 | 33 | 49
Insomnia (Psychiatric disorders) | 26 | 21 | 42
Cough (Respiratory, thoracic and mediastinal disorders) | 41 | 47 | 65
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 18 | 10 | 24
Rash (Skin and subcutaneous tissue disorders) | 28 | 29 | 40
Hypertension (Vascular disorders) | 14 | 26 | 39

LIMITATIONS AND CAVEATS:
10 participants from a single study site were excluded from Intent-to-Treat (ITT) Analysis Set due to critical and multiple protocol violations (elvitegravir arm: n = 3; raltegravir arm: n = 7).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years